CLINICAL TRIAL: NCT00794677
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Period, Crossover Study to Evaluate the Effects of Ezetimibe on the Plasma Appearance of 7-Ketocholesterol After an Oral Bolus in Patients With Primary Hypercholesterolemia
Brief Title: Effects of Ezetimibe on the Absorption of Oxidized Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Merck Schering-Plough (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MM6997
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Oxysterol; Ezetimibe; Zetia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo medication will be taken orally once daily in the morning on rising either during the first intervention period or the second intervention period. Single-blind ezetimibe placebo will be taken during the Run-In Period. Patients will be issued one bottle containing either active drug or placebo for each treatment period.
  Interventions: Drug: placebo
- ezetimibe (Experimental): 10 mg medication will be taken orally once daily in the morning on rising either during the first intervention period or the second intervention period. Single-blind ezetimibe placebo will be taken during the Run-In Period. Patients will be issued one bottle containing either active drug or placebo for each treatment period.
  Interventions: Drug: ezetimibe

INTERVENTIONS:
Drug: ezetimibe — Blinded study medication (ezetimibe 10 mg in tablet form) will be taken orally once daily in the morning on rising. Single-blind ezetimibe placebo will be taken during the Run-In Period. Patients will be issued one bottle containing either active drug or placebo for each treatment period.
  Other Names: Zetia
  Arms: ezetimibe
Drug: placebo — Blinded study medication (matched placebo) will be taken orally once daily in the morning on rising. Single-blind ezetimibe placebo will be taken during the Run-In Period. Patients will be issued one bottle containing either active drug or placebo for each treatment period.
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to test the effects of Zetia™ (ezetimibe) 10 milligrams (mg) on the absorption of oxysterol into the blood following a meal containing oxysterol.

DETAILED DESCRIPTION:
There are a number of cholesterol-lowering drugs available that can lower blood cholesterol to a healthier level. Zetia™ (ezetimibe) 10 mg is available by prescription for the treatment of high cholesterol. While Zetia has been shown to inhibit the absorption of dietary cholesterol into the bloodstream, its effects on oxysterol absorption from the diet have not been completely evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant or lactating and is highly unlikely to conceive
* Body Mass Index (BMI) between 20-30 kilograms per meter squared (kg/m2) inclusive.
* Body weight, as reported by patient, stable (±2 kg) for >6 weeks
* Plasma low density lipoprotein cholesterol (LDL-C) between 130 and 180 milligrams per deciliter (mg/dL) inclusive. Note: One retest allowed.
* Triglyceride (TG) concentrations ≤150 mg/dL. Note: One retest allowed.
* Fasting blood glucose <110 mg/dL and hemoglobin A1c (HbA1C) ≤ 6 percent at Visit 1. Note: One retest allowed.
* Liver transaminases (ALT, AST) ≤1.5 x upper limit of normal (ULN) and no active liver disease. Note: One retest allowed.
* Creatine Phosphokinase (CPK) ≤2x ULN. Note: One retest allowed.
* Willingness to maintain a stable diet for the duration of the study.
* Can understand and comply with study procedures and signs a written informed consent.
* Patient is ≥80 precent compliant with dosing during Placebo Run-In Period or, in the opinion of the investigator, is able to maintain ≥80 percent therapy compliance during the active treatment period of the study.

Exclusion Criteria:

* Lipid-lowering therapy and replacement of this therapy with study medication is considered inappropriate by the investigator.
* Consumes an average of more than 2 alcoholic drinks per day.
* Smokes.
* Currently engages in a vigorous exercise regimen or intensive exercise bouts >4x per month.
* Treated with any other investigational drug within 30 days of Visit 1.
* Hypersensitivity or intolerance to ezetimibe or any component of this medication.
* Any condition or situation which poses a risk to the patient or interfere with participation in the study.
* Congestive heart failure.
* Uncontrolled cardiac arrhythmias.
* History of myocardial infarction, stroke, or any other clinical manifestation of coronary, cerebral, or peripheral vascular disease.
* Uncontrolled hypertension
* Impaired renal function, nephrotic syndrome or other clinically significant renal disease at Visit 1.
* Active or chronic hepatobiliary or hepatic disease.
* History of irritable bowel syndrome, ileal bypass, gastric bypass or any gastrointestinal disorder/condition associated with malabsorption.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins.
* Type I or Type II diabetes mellitus.
* Disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Human Immunodeficiency Virus (HIV) positive.
* History of cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of uncontrolled psychiatric illness or drug/alcohol abuse within the past 5 years. Individuals with psychiatric illness adequately controlled and stable on pharmacotherapy may be enrolled at the discretion of the investigator.
* Lipid-lowering agents taken within 6 weeks and fibrates taken within 8 weeks prior to visit 3.
* Cardiovascular medications are acceptable provided the patient has been on a stable regimen for at least 6 weeks prior to Visit 3 and indicates a willingness to continue the stable regimen for the duration of the study.
* Supplementation with antioxidants beyond a standard multivitamin for the duration of the study.
* Psyllium, other fiber-based laxatives, and/or over the counter (OTC) therapies known to affect serum lipid levels taken within 6 weeks of Visit 3.
* Female patients receiving hormone replacement therapy, any estrogen antagonist/agonist or hormonal contraceptives.
* Treatment with cyclosporine except for ophthalmic indication
* Anti-obesity medications such as orlistat or sibutramine taken within 3 months prior to Visit 1.
* Therapeutic doses of systemic corticosteroids except inhaled steroid therapy (for example, Pulmicort®) maintained on a stable dosing regimen for at least 6 weeks prior to randomization (Visit 3) and throughout the duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in 2007 through search of a clinical research center database, mailings to homes, and posted flyers in the Berkeley, California area.
Pre-assignment Details: 55 participants screened; 29 excluded because they did not meet inclusion criteria
Groups:
- Placebo First: Placebo once daily in first intervention period and ezetimibe (10 mg/day) in second intervention period
- Ezetimibe First: Ezetimibe (10 mg/day) once daily in the first intervention period and placebo once daily in the second intervention period
Period: First Intervention
Arm/Group | Placebo First | Ezetimibe First
Started | 13 | 13
Completed | 11 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Placebo First | Ezetimibe First
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ezetimibe: Ezetimibe (10 mg/day) once daily received as the first or second intervention
- Placebo: Placebo once daily received as the first or second intervention
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.05 (7.54) | 50.09 (14.28) | 50.99 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24.0

OUTCOME MEASURES:

1. Primary Outcome: Log[Area-under-the-plasma-concentration-curve(AUC) 0-8 Hours 7-ketocholesterol] After an Oral Bolus
Description: Log of Area-under-the-plasma-concentration curve (AUC 0-8hrs) of 7-ketocholesterol after an oral bolus in patients with primary hypercholesterolemia after treatment with ezetimibe versus placebo
Time Frame: 6 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: Log(mg*hr/dl)
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
Log(mg*hr/dl) | 1.925 (0.166) | 2.177 (0.142)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Statistical significance was determined for a standard two-period crossover design using JMP software (Version 5.0, SAS Institute. Cary, NC); Test type: Superiority or Other; p = 0.03, ANOVA; Mean Difference (Final Values) = -0.252, Standard Error of Mean 0.112

2. Secondary Outcome: Log(Maximal Plasma Concentration (Cmax) of 7-ketocholesterol) After an Oral Bolus
Description: Log Cmax of 7 ketocholesterol after an oral bolus in patients with primary hypercholesterolemia.
Time Frame: 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: Log(mg/dl)
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
Log(mg/dl) | 0.973 (0.156) | 1.246 (0.133)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = -0.273, Standard Error of Mean 0.102

3. Other Pre Specified Outcome: Log(Fasting Plasma Levels of Diet-derived Oxysterols (7-ketocholesterol))
Time Frame: 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: Log(mg/dl)
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
Log(mg/dl) | -1.119 (0.124) | -1.070 (0.107)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.60, ANOVA; Mean Difference (Final Values) = -0.048, Standard Error of Mean 0.089

4. Other Pre Specified Outcome: Log (AUC of Plasma Total Cholesterol) After an Oral Bolus
Description: Area under the curve (AUC) calculated over 8 hours
Time Frame: 6 weeks
Population: Per protocol, restricted to changes that were nonnegative because there is no log for a negative number
Measure: Mean (Standard Error); unit: Log(mg*hr/dl)
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 9 | 9
Log(mg*hr/dl) | 2.928 (0.213) | 2.719 (0.346)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.67, ANOVA; Mean Difference (Final Values) = 0.209, Standard Error of Mean 0.470

5. Other Pre Specified Outcome: Log (AUC of Plasma Triglyceride) After an Oral Bolus
Description: Area under the curve (AUC) calculated over 8 hours
Time Frame: 6 weeks
Population: Per protocol, one subject eliminated because the AUC was negative and cannot be log transformed
Measure: Mean (Standard Error); unit: Log(mg*hr/dl)
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 23 | 23
Log(mg*hr/dl) | 4.894 (0.139) | 5.044 (0.126)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.30, ANOVA; Mean Difference (Final Values) = -0.150, Standard Error of Mean 0.140

6. Other Pre Specified Outcome: Percent Change of Fasting Apolipoprotein B From Baseline
Description: Change = [(Week 6 - baseline)/baseline value *100]
Time Frame: Baseline (placebo run-in) and 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
percent change from baseline | -17.990 (1.648) | -2.577 (2.113)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Net) = -15.412, Standard Error of Mean 1.569

7. Other Pre Specified Outcome: Percent Change of Fasting Low Density Lipoprotein Cholesterol From Baseline
Description: Change = [(Week 6 - baseline)/baseline value *100]
Time Frame: Baseline (placebo run-in) and 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
percent change from baseline | -22.891 (2.497) | -1.045 (2.454)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.0000001, ANOVA; Mean Difference (Net) = -21.846, Standard Error of Mean 2.866

8. Other Pre Specified Outcome: Percent Change in Fasting High Density Lipoprotein Cholesterol
Description: Change = [(Week 6 - baseline)/baseline value *100]
Time Frame: Baseline (placebo run-in) and 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
percent change from baseline | -1.936 (2.134) | -7.333 (1.860)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p = 0.009, ANOVA; Mean Difference (Net) = 5.397, Standard Error of Mean 1.893

9. Other Pre Specified Outcome: Percent Change of Fasting Non-high Density Lipoprotein Cholesterol From Baseline
Description: Change = [(Week 6 - baseline)/baseline value *100]
Time Frame: Baseline (placebo run-in) and 6 weeks
Population: Per protocol
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 24 | 24
percent change from baseline | -22.675 (2.326) | -1.322 (1.871)
Statistical Analysis 1: Comparison: Ezetimibe vs Placebo; Test type: Superiority or Other; p < 0.0000001, ANOVA; Mean Difference (Net) = -21.353, Standard Error of Mean 2.220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No